CLINICAL TRIAL: NCT03132246
Title: Early Determination of Biofilm Formation on Orthopaedic Devices
Brief Title: MICRO Study: Detecting Bacterial Infections Related to Orthopaedic Surgical Implants
Acronym: MICRO
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert O'Toole, Head of the UM SOM's Division of Orthopaedic Traumatology and Chief of Orthopaedic Traumatology and CHief of Orthopaedics for the University of Maryland Medical Center's (UMMS) R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Other Study IDs: HP-00055743
Record Dates: First submitted 2017-04-07; First posted 2017-04-27 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Open Reduction and Internal Fixation of Extremity Fractures
Keywords: Methicillin-resistant Staphylococcus aureus (MRSA); Infection; Biofilm Assay
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Infected: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. Each patient enrolled in the study provided 1-3 blood samples. These blood samples were tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.
  Patients were enrolled if presented as high risk but later separated into the Infected Group or the Not Infected Group based on whether or not they went on to develop an infection post surgery. All patients in this group went on to develop an infection.
  Interventions: Diagnostic Test: Blood draws
- Not Infected: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. Each patient enrolled in the study provided 1-3 blood samples. These blood samples were tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.
  Patients were enrolled if presented as high risk but later separated into the Infected Group or the Not Infected Group based on whether or not they went on to develop an infection post surgery. All patients in this group did not go on to develop an infection.
  Interventions: Diagnostic Test: Blood draws

INTERVENTIONS:
Diagnostic Test: Blood draws — The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.

SUMMARY:
A prospective trial conducted at Shock Trauma of patients between 18 years of age and older who have sustained a fracture with metal implanted. The investigators will be collecting between 1-3 routine blood draws for the purpose of laboratory analysis to assess biofilm growth. Patients may be infected or non-infected at the time of blood draw; they will be selected at random for purposes of this study. All patients will be followed as standard of care by their treating physician for all their follow up visits.

DETAILED DESCRIPTION:
Surgical site infection in the orthopaedic surgery population is a significant public health issue. Wound infections result in both increased length of hospital stay and total cost of care.

Surgical site infection (SSI) is the most common preventable adverse outcome after a major operation. The economic costs to the US healthcare system are enormous estimated to be in excess of $1.8 billion per year. For patients who develop an SSI, the cost may be even higher with length of stay and risk of death doubled. Thus the benefits of any intervention decreasing the risk of SSI are very tangible.

A biofilm is a layer of bacteria that adheres to a surface; in Orthopaedics, this often means adherence to implanted metal after fracture surgery. The test that has been designed by one of the investigators on the study has been shown in an animal model to detect the formation of a biofilm up to 1 month prior to clinical detection. Having a blood assay such as this would allow earlier antibiotics and potentially prevent the need for further surgeries to remove metal implants and clean out the biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Previous fracture fixation with an implant (intramedullary nail, plate, screws), or joint revisions, or periprosthetic fracture, or admitted from orthopaedic trauma clinic due to infection, or inpatient with a known infection.
* English speaking

Exclusion Criteria:

* Patients with planned follow-up at another medical center
* Patient lives outside of the hospital catchment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert V O'Toole, MD, Principal Investigator — University of Maryland, College Park; Mark Shirtliff, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Shock Trauma Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Prabhakara R, Harro JM, Leid JG, Harris M, Shirtliff ME. Murine immune response to a chronic Staphylococcus aureus biofilm infection. Infect Immun. 2011 Apr;79(4):1789-96. doi: 10.1128/IAI.01386-10. Epub 2011 Jan 31. PMID 21282411

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were enrolled if presented as high risk but later separated into the Infected Group or the Not Infected Group based on whether or not they went on to develop an infection post surgery. Group assignment is unknown for patients that did not complete the study and therefore groups are combined for reporting overall study numbers.
Groups:
- Enrolled: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. Each patient enrolled in the study provided 1-3 blood samples. These blood samples were tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.
  Patients were enrolled if presented as high risk but later separated into the Infected Group or the Not Infected Group based on whether or not they went on to develop an infection post surgery. Group assignment is unknown for patients that did not complete the study and therefore groups are combined for reporting overall study numbers.
Period: Overall Study
Arm/Group | Enrolled
Started | 260
Completed | 156
Not Completed | 104

BASELINE CHARACTERISTICS:
Population: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation.
Groups:
- Infected: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. All patients in this arm went on to develop an infection. Each patient enrolled in the study provides blood samples up to 10 times. These blood samples are to be tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  Blood draw: The only intervention patients experience is a non-standard of care blood draw. The blood is then tested in a basic science laboratory.
- Not Infected: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. All patients in this arm did not go on to develop an infection. Each patient enrolled in the study provides blood samples up to 10 times. These blood samples are to be tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  Blood draw: The only intervention patients experience is a non-standard of care blood draw. The blood is then tested in a basic science laboratory.
- Total: Total of all reporting groups
Arm/Group | Infected | Not Infected | Total
Number analyzed (Participants) | 20 | 136 | 156
Age, Continuous [Mean (Full Range); unit: years] | 45 [18 to 81] | 44 [22 to 62] | 44 [18 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 51 | 56
  Male | 15 | 85 | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Full Range); unit: kg/m2] | 27 [18 to 45] | 28 [17 to 49] | 28 [17 to 49]
Smoker [Count of Participants; unit: Participants] | 12 | 55 | 67
Follow up [Mean (Full Range); unit: months] | 58 [18 to 121] | 28 [18 to 58] | 43 [18 to 121]
Time to Infection [Mean (Full Range); unit: months] — Population: This measure is only valid for infection patients.
  months
    number analyzed (Participants) | 20 | 0 | 20
    (all) | 11 [1 to 90] |  | 11 [1 to 90]
Open Fracture [Count of Participants; unit: Participants] | 8 | 51 | 59
Closed Fractures [Count of Participants; unit: Participants] | 12 | 85 | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Blood Samples With High Levels of Absorbance Via ELISA for Patients (Greater Than 1.5 Ratio Compared to Control Human Serum)
Description: A high level of absorbance via ELISA (greater than 1.5 ratio compared to control human serum) is a positive test result. The rate of not infected patient samples that return positive will demonstrate the false positive rate of the test.
Time Frame: 1 year of clinical follow-up
Population: One to three blood sample tests were taken for each participant prior to the one-year post-operative clinical follow-up. Clinical cultures will also be monitored for the one-year post-operative period and compared to the blood sample test results to determine if the test is able to identify patients with positive staphylococcal infection cultures.
Measure: Count of Units; unit: blood draw samples
Units Other Than Participants: blood draw samples
Arm/Group | Infected | Not Infected
Number analyzed (Participants) | 20 | 136
Number analyzed (blood draw samples) | 52 | 145
blood draw samples | 48 | 53

2. Secondary Outcome: Number of Blood Samples With Low Levels of Absorbance Via ELISA for Patients (Greater Than 1.5 Ratio Compared to Control Human Serum)
Description: A low level of absorbance via ELISA (greater than 1.5 ratio compared to control human serum) is a negative test result. The rate of infected patient samples that return negative will demonstrate the false negative rate of the test.
Time Frame: 1 year of clinical follow-up
Population: as for outcome 1
Measure: Count of Units; unit: blood draw samples
Units Other Than Participants: blood draw samples
Arm/Group | Infected | Not Infected
Number analyzed (Participants) | 20 | 136
Number analyzed (blood draw samples) | 52 | 145
blood draw samples | 4 | 92

ADVERSE EVENTS:
Time Frame: 3 months - 1 year depending on if the patient experienced a clinical culture return of staphylococcal-positive
Groups:
- Unmasked Non-completers: Trauma patients that were considered at risk for infection after fracture fixation. Inclusion criteria included open fractures, proximal tibia fractures, pilon fractures, and calcaneus fractures treated with surgical fixation. Each patient enrolled in the study provided 1-3 blood samples. These blood samples were tested using basic science techniques to determine the level of exposure to a staphylococcal biofilm each patient has experienced over a period of time.
  The only intervention patients experience are non-standard of care blood draws. The blood is then tested in a basic science laboratory.
  Patients were enrolled if presented as high risk but later separated into the Infected Group or the Not Infected Group based on whether or not they went on to develop an infection post surgery. Group assignment is unknown for patients that did not complete the study and therefore this group is representative of those patients that were enrolled but did not complete the study.
Arm/Group | Unmasked Non-completers | Infected | Not Infected
All-Cause Mortality (participants affected / at risk) | 0/104 | 1/20 | 3/136
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/20 | 0/136
Other Adverse Events (participants affected / at risk) | 0/104 | 0/20 | 0/136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT03132246/Prot_SAP_000.pdf